CLINICAL TRIAL: NCT03008772
Title: REWARDS-In-stent Restenosis
Brief Title: REWARDS- In-stent Restenosis
Status: Withdrawn | Type: Observational
Why Stopped: Not funded
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: REWARDS-ISR
Record Dates: First submitted 2016-12-21; First posted 2017-01-02 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: In-Stent Coronary Artery Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PCI with Commercially available DES: Patients who have undergone PCI and received a commercially available drug eluting stent
- Stent Types: the stent types for angina classification at follow up

SUMMARY:
To define the long-term incidence and frequency of ISR follow DES implantation. Compare the clinical presentation, treatment and intervention success among de novo coronary artery stenosis and DES ISR.

Compare short- and long-term outcomes of de novo coronary artery stenosis and DES ISR, assessed by incidence of mortality, MACE, MI, and TLR/TVR at index hospitalization, 30 days, 6 months, 1 year, 3 years, and 5 years, if available.

DETAILED DESCRIPTION:
Drug-eluting coronary stents (DES) significantly reduced the rate of neointimal hyperplasia and in-stent restenosis (ISR) compared to bare metal stents (BMS) for the treatment of coronary artery disease. In addition, the continued evolution in scaffold and polymer design with concomitant improvements in antiplatelet therapy has improved the rates of late and very late stent thrombosis. However, despite novel metal scaffold technology, increasing operator experience, and improvement in adjunctive implantation techniques, the incidence of ISR in durable-polymer DES remains a problem, with 1-year rates as high as 12 to 15%.

The outcomes associated with ISR highlight the fact that this is by no means a benign process and studies report MI rates as high as 19.4% with one study demonstrating a total rate of death or nonfatal MI of 3.5%. In addition, ISR presenting as acute coronary syndrome (ACS) has an independent effect on major adverse cardiac events. The emergence of fully bioresorbable vascular scaffolds (BVS) has provided an exciting alternative to combat the long-term structural and functional effects on the coronary vessel seen with implantation of a permanent metal scaffold, regardless of the drug coating. Initial studies have demonstrated the non-inferiority of BVS compared to contemporary DES in regards to death, MI, and MACE. In addition, intravascular imaging has confirmed complete resorbtion of the BVS by 3 years time. The long-term benefits of such technology have yet to be fully assessed. However, based on literature outlining the complicated course of ISR in short-term and that seen in the bare metal stent era, it is projected that complete resorbtion of the vascular scaffold should improve long-term outcomes of patients with ischemic heart disease.

Currently, the clinical presentation, incidence, and outcomes of ISR in contemporary DES are not completely understood. The goal of this particular study is to retrospectively evaluate the long-term impact of ISR over a 10-year period in current contemporary DES. The data can be compared to de novo coronary artery lesions with similar characteristics and complexity to highlight the significant differences in the clinical course of each disease. Ultimately, the investigators will hopefully demonstrate the need for improvement in this arena, which the BVS will potentially provide.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, > 18 years of age,
* Patients who received at least one (1) commercially available Drug Eluting Stent

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study subjects will be identified retrospectively. Patients who have undergone PCI and received a commercially available drug eluting stent as listed above. These patients will be compared between the stent types for angina classification at follow up.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Instent Restenosis | Up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No